CLINICAL TRIAL: NCT02928016
Title: Effectiveness of the Carbohydrate Counting Method on Postprandial Glucose Concentrations After Consumption of Mixed Meals in Adults With Type 1 Diabetes
Brief Title: Effectiveness of Carbohydrate Counting Method With Mixed Meals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agricultural University of Athens (Other)
Collaborators: Harokopio University (Other)
Responsible Party: Principal Investigator, Aimilia Papakonstantinou, Lecturer in Nutrition and Metabolism Unit of Human Nutrition Dept of Food Science and Human Nutrition Agricultural University Of Athens, Agricultural University of Athens
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: HRBD 11th Session 6/4/2014 NHA
Record Dates: First submitted 2016-10-06; First posted 2016-10-07 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Type 1 Diabetes
Keywords: carbohydrate counting method; protein; fat; glucose; type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Platelet Glycoprotein IV Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Mixed meal 1 (Experimental): 20 adults with type 1 diabetes (T1DM) on intensive insulin treatment and glycated haemoglobin (HbA1c) <10% consumed three ready-made standardised mixed meals (a dish made with thick pasta, minced meat and béchamel sauce, grilled chicken with vegetables and baked giant beans) with and without the addition of 11 ml of extra virgin olive oil within 20 minutes. No other food or drink (except for water) were consumed until the end of the trial period (total duration 195 minutes). Participants consumed all meals in random order during 6 consecutive visits with one week wash-out period in between visits.
  Interventions: Other: Mixed meal 1
- Mixed meal 2 (Experimental): 20 adults with type 1 diabetes (T1DM) on intensive insulin treatment and glycated haemoglobin (HbA1c) <10% consumed three ready-made standardised mixed meals (a dish made with thick pasta, minced meat and béchamel sauce, grilled chicken with vegetables and baked giant beans) with and without the addition of 11 ml of extra virgin olive oil within 20 minutes. No other food or drink (except for water) were consumed until the end of the trial period (total duration 195 minutes). Participants consumed all meals in random order during 6 consecutive visits with one week wash-out period in between visits.
  Interventions: Other: Mixed meal 2
- Mixed meal 3 (Experimental): 20 adults with type 1 diabetes (T1DM) on intensive insulin treatment and glycated haemoglobin (HbA1c) <10% consumed three ready-made standardised mixed meals (a dish made with thick pasta, minced meat and béchamel sauce, grilled chicken with vegetables and baked giant beans) with and without the addition of 11 ml of extra virgin olive oil within 20 minutes. No other food or drink (except for water) were consumed until the end of the trial period (total duration 195 minutes). Participants consumed all meals in random order during 6 consecutive visits with one week wash-out period in between visits.
  Interventions: Other: Mixed meal 3
- Mixed meal 4 (Experimental): 20 adults with type 1 diabetes (T1DM) on intensive insulin treatment and glycated haemoglobin (HbA1c) <10% consumed three ready-made standardised mixed meals (a dish made with thick pasta, minced meat and béchamel sauce, grilled chicken with vegetables and baked giant beans) with and without the addition of 11 ml of extra virgin olive oil within 20 minutes. No other food or drink (except for water) were consumed until the end of the trial period (total duration 195 minutes). Participants consumed all meals in random order during 6 consecutive visits with one week wash-out period in between visits.
  Interventions: Other: Mixed meal 4
- Mixed meal 5 (Experimental): 20 adults with type 1 diabetes (T1DM) on intensive insulin treatment and glycated haemoglobin (HbA1c) <10% consumed three ready-made standardised mixed meals (a dish made with thick pasta, minced meat and béchamel sauce, grilled chicken with vegetables and baked giant beans) with and without the addition of 11 ml of extra virgin olive oil within 20 minutes. No other food or drink (except for water) were consumed until the end of the trial period (total duration 195 minutes). Participants consumed all meals in random order during 6 consecutive visits with one week wash-out period in between visits.
  Interventions: Other: Mixed meal 5
- Mixed meal 6 (Experimental): 20 adults with type 1 diabetes (T1DM) on intensive insulin treatment and glycated haemoglobin (HbA1c) <10% consumed three ready-made standardised mixed meals (a dish made with thick pasta, minced meat and béchamel sauce, grilled chicken with vegetables and baked giant beans) with and without the addition of 11 ml of extra virgin olive oil within 20 minutes. No other food or drink (except for water) were consumed until the end of the trial period (total duration 195 minutes). Participants consumed all meals in random order during 6 consecutive visits with one week wash-out period in between visits.
  Interventions: Other: Mixed meal 6

INTERVENTIONS:
Other: Mixed meal 1 — 20 adults with type 1 diabetes (T1DM) on intensive insulin treatment consumed a dish made with thick pasta, minced meat and béchamel sauce and 20 g kalamata olives. The meal provided 794 kcal and contained approximately 500 kcal from protein and fat. Insulin requirements for the test meal were calculated based on the carbohydrate content of the dish according to the personalised carbohydrate to insulin ratio.
  Arms: Mixed meal 1
Other: Mixed meal 2 — 20 adults with type 1 diabetes (T1DM) on intensive insulin treatment consumed grilled chicken with vegetables.The meal provided 399 kcal and contained approximately 300 kcal from protein and fat. Insulin requirements for the test meal were calculated based on the carbohydrate content of the dish according to the personalised carbohydrate to insulin ratio.
  Arms: Mixed meal 2
Other: Mixed meal 3 — 20 adults with type 1 diabetes (T1DM) on intensive insulin treatment consumed baked giant beans and 20g kalamata olives. The meal provided 502 kcal and contained approximately 300 kcal from protein and fat. Insulin requirements for the test meal were calculated based on the carbohydrate content of the dish according to the personalised carbohydrate to insulin ratio.
  Arms: Mixed meal 3
Other: Mixed meal 4 — 20 adults with type 1 diabetes (T1DM) on intensive insulin treatment consumed a dish made with thick pasta, minced meat and béchamel sauce and 20 g kalamata olives and 11 ml extra virgin olive oil. The meal provided 893 kcal and contained approximately 600 kcal from protein and fat. Insulin requirements for the test meal were calculated based on the carbohydrate content of the dish according to the personalised carbohydrate to insulin ratio.
  Arms: Mixed meal 4
Other: Mixed meal 5 — 20 adults with type 1 diabetes (T1DM) on intensive insulin treatment consumed grilled chicken with vegetables and 11 ml extra virgin olive oil. The meal provided 497 kcal and contained approximately 300 kcal from protein and fat. Insulin requirements for the test meal were calculated based on the carbohydrate content of the dish according to the personalised carbohydrate to insulin ratio.
  Arms: Mixed meal 5
Other: Mixed meal 6 — 20 adults with type 1 diabetes (T1DM) on intensive insulin treatment consumed baked giant beans and 20 g kalamata olives and 11 ml extra virgin olive oil. The meal provided 601 kcal and contained approximately 400 kcal from protein and fat. Insulin requirements for the test meal were calculated based on the carbohydrate content of the dish according to the personalised carbohydrate to insulin ratio.
  Arms: Mixed meal 6

SUMMARY:
In a randomized, cross-over designed study, the investigators examined the effectiveness of the carbohydrate counting method after consumption of mixed meals typical of the Greek cuisine with various protein and fat contents in a sample of people with type 1 diabetes (DM1). The investigators also tried to further explore the effects of additional extra virgin olive oil (11 ml) on the glycemic response.

DETAILED DESCRIPTION:
A total of 20 adults with type 1 diabetes on intensive insulin therapy consumed three mixed meals at noon between 1200 and 1300 hours, with and without the addition of 11 ml extra virgin oil, in random order. One week before entering the study, participants kept a detailed 7-day weighed food record with fingerprick blood glucose measurements pre-and-2hour post-meals for calculation of their carbohydrate (g) to insulin (units) ratio. Moreover, the individual correction factor was calculated. Thereafter, insulin requirements for the test meals were calculated based on the carbohydrate content of each dish and according to the personalised carbohydrate to insulin ratio. Postprandial glycemia was measured in capillary blood glucose samples at 30min intervals over 195min. For 24hr before each testing session, participants were asked to refrain from the consumption of alcohol and to maintain their usual physical activity pattern. On the day of testing, subjects were asked to consume their usual breakfast and abstain from food for at least 2 hours before their appointment. If blood glucose was >7.2 mmol/l at 1200, insulin was administered based on the individualised correction factor. If blood glucose was >10 mmol/l at the beginning of the testing session, insulin was administered to correct it and the subject was asked to return on another day. if hypoglycaemia occurred (defined as blood glucose level <3.8 mmol/l), the test session was stopped, the event was recorded and the patient treated appropriately. The on target 2hour postprandial blood glucose level was set between 3.9 and 10 mmol/l. Anthropometric measurements (body weight, waist and hip circumferences) were performed at every visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 1 diabetes
* Intensive insulin therapy
* HbA1c < 10%
* >2 years with diabetes

Exclusion Criteria:

* Food allergies
* Diabetic neuropathy
* Kidney disease
* Hematological disturbances
* Liver disease
* Uncontrolled hypo- or hyperthyroidism
* Arrhythmia
* Heart disease
* Cancer
* Serious mental illness

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2014-09; Primary Completion 2015-04 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Capillary blood glucose | 195 minutes
  Clinically useful change in capillary blood glucose, defined as the restoration of glucose within normal limits during the first two hours and until the end of the trial

CONTACTS AND LOCATIONS:
Overall Officials: Aimilia Papakonstantinou, PhD, Principal Investigator — Agricultural University of Athens

IPD SHARING:
Plan to Share IPD: No